CLINICAL TRIAL: NCT04300712
Title: Partnerships Between Schools and Public Mental Health Departments: Investigation of Multi-professional Interventions for Children Aged 3 to 8 With Mental Health Issues (Parpsych-Ed).
Acronym: Parpsych-Ed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GCS pour la recherche et la formation en sante mentale (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Parpsych-Ed_2018
Record Dates: First submitted 2019-05-10; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: School Difficulties Associated With Mental Health Problems
Keywords: mental health; children psychiatry; school difficulties; psychosocial interventions
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tracking of the children with difficulties (Other): All parents and teachers will respond to the questionnaires and the beginning and end of school year which is not done in the routine for tracking the children in difficulty.
  Interventions: Behavioral: Questionnaires at the start and end of the school year

INTERVENTIONS:
Behavioral: Questionnaires at the start and end of the school year — Interventions will be proposed to children identified in a worrisome situation. The Strengths and Difficulties. Questionnaire will be used by teachers to score these situations. The recognition process of mental health problem and need continue with responses. Responses are supporting a graduated response process in school and facilitating external support when needed (mental health services, community supports). Early intervention is one of all responses, which involve caregivers. Responses to worrisome situations aim to improve schooling conditions, to acknowledge mental health problems or condition and the health services need for children. To evaluate the intervention, the impact supplement of SDQ and the follow-up questions will be used by the teachers and the parents of children who benefit of the intervention. The interventions will be experimented during year 2020-21. Children might benefit of them from several weeks to one year, according to their need.
  Other Names: Questionnaires at the start and end of the school year completed by teachers and directors; Questionnaire before and after intervention completed by teachers and parents.; Questionnaires during and after the intervention, completed by public mental health professionals

SUMMARY:
Local partnerships between schools (preschool and elementary) and mental health public services are implemented in seven sites in France. They aim to improve recognition of difficulties related to mental health problems and to provide interventions to 3 to 8 years-old pupils in need. Our hypothesis that these local partnerships and interventions enhance the role of school in supporting good mental health and wellbeing of all children and the trajectories of children with mental health service needs. Theses also facilitate community support. One of them, early-interventions involve caregivers. Our objective is to enhance knowledge of the unmet mental healthcare need at school and to explore for whom, in which local context and how partnerships and early intervention work.

DETAILED DESCRIPTION:
Teachers are legitimately concerned about children that encounter mental health problems. Mental healthcare might be indicated. Because of internal and external barriers of treatment, they could remain inaccessible for many children in need. School staff should not try to diagnose conditions. However, collaborative interventions delivered by school and mental healthcare staffs in association with other stakeholders as parents and associations should ensure clear systems and processes in place for identifying possible mental health problems and support children and their parents. Local partnership and early interventions will be elaborated within focus groups bringing together all stakeholders and will be experimented in 7 French sites (preschool, primary school and local public health service) thereafter. These complex interventions will be evaluated through mixed-methods including qualitative case studies and a pragmatic trial. This feasibility study will produce a set of findings that will permit to argue conceptual framework of partnership and early intervention, to provide guidelines to implement these in France considering children needs, local context, all stakeholders acceptance and public health efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Attending pre- and elementary schools involved in the ParpsychEd partnerships.

Exclusion Criteria:

* Absence of parents and/or child consent.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
number of 3 to 8 years old children identified with mental health services need | 24 months
  Evolution of the number of 3 to 8 years old children identified with mental health services

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | 12 months
  Changes in the impact supplement and the follow-up questions - parents and teachers
Healthcare access, barriers to treatment, intervention acceptance | 12 months
  Healthcare access, barriers to treatment, intervention acceptance
Parent refusal rate to let their child benefit of all responses | 12 months
  Parent refusal rate to let their child benefit of all responses
Parent refusal rate to let their child benefit of the early intervention | 12 months
  Parent refusal rate to let their child benefit of the early intervention
Parents refusal rate to plan appointment in public health services as indicated after the intervention | 18 months
  Parents refusal rate to plan appointment in public health services as indicated after the intervention
Mental health and mental health services representation and use | 18 months
  Changes in the mental health representations of parents, teachers and others professionnals

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Roelandt, MD, Study Director — French World Health Organization Collaborating Centre for Research and Training in Mental Health; Sandrine Bonneton, MD, Principal Investigator — French World Health Organization Collaborating Centre for Research and Training in Mental Health
Locations (7):
- France (7):
  - EPSM Barthélémy Durand, Grigny, Essone
  - EPSM de Guadeloupe, Saint-Claude, Guadeloupe
  - EPSM Val de Lys, La Couture, Pas De Calais
  - EPSM Val de Lys, Vieille Chapelle, Pas De Calais
  - Centre Hospitalier Sainte Anne, Paris
  - Fondation Bon Sauveur de la Manche, Picauville
  - Centre Hospitalier de Saint Denis, Saint-Denis

IPD SHARING:
Plan to Share IPD: Undecided